CLINICAL TRIAL: NCT00137709
Title: Hormone Profiles in Adults Treated With Valproate vs. Lamotrigine Monotherapy for Newly Diagnosed Epilepsy: A Prospective Randomised Study
Brief Title: Hormone Profiles in Adults With Newly Diagnosed Epilepsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2004.399
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Epilepsy
Keywords: epilepsy; hormone
MeSH Terms: conditions — Epilepsy | interventions — Valproic Acid; Lamotrigine

INTERVENTIONS:
Drug: Sodium valproate — Week 1 & 2 - 200mg twice daily Week 3 onwards - 400mg twice daily
Drug: Lamotrigine — Week 1 - 25mg mane Week 2 - 25mg twice daily Week 3 - 25mg mane, 50mg nocte Week 4 onwards - 50mg twice daily

SUMMARY:
Both sodium valproate and lamotrigine are currently used in the treatment of newly diagnosed epilepsy. Although they appear to have similar efficacy, they have different side effects, which have not been well studied. This study aims to compare one particular aspect of their possible side effects, namely whether they affect certain hormonal functions.

DETAILED DESCRIPTION:
Sodium valproate is an established antiepileptic drug used against a broad range of seizure types. Lamotrigine, a newer antiepileptic drug available since late 1980s, has a similar range of action and is approved as first-line treatment for epilepsy in the United States and many European countries as well as in Hong Kong. Recently, concern has been raised over the association between valproate treatment and polycystic ovarian syndrome, a condition characterised by multiple cysts in the ovaries in women and a range of hormonal and metabolic disturbances. Cross-sectional studies from Finland suggest that up to 40% of women treated with valproate have polycystic ovaries. Lamotrigine substitution for valproate has been reported to normalise these parameters in some patients. Elevated serum insulin and androgen levels have also been reported in over 50% of male patients taking valproate for epilepsy. However, such high incidence of hormonal abnormalities associated with valproate treatment has not been reproduced in studies conducted in other western populations. No similar studies in Chinese patients have been reported. In addition, these cross-sectional studies suffer from many potential confounding factors, such as previous treatment with other antiepileptic drugs, variation in duration of treatment, thus limiting the ability to establish a causal relationship.

This phase IV study aims to examine whether valproate treatment is associated with hormonal abnormalities in Chinese epilepsy patients. Newly diagnosed patients will be randomised to receive valproate or lamotrigine and their hormonal profiles measured prospectively for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 15 and 55
* Ethnically Chinese
* Newly diagnosed epilepsy requiring antiepileptic drug treatment; or patients previously treated with antiepileptic drugs but have withdrawn from medication for at least 1 year, and now require resumption of antiepileptic drug therapy due to seizure relapse.

Exclusion Criteria:

* Post-menopausal women.
* Pregnant women.
* Women who have undergone oophorectomy.
* Women taking or have taken oral contraceptive pills in the previous 3 months.
* Women diagnosed with or suspected to have polycystic ovarian syndrome.
* Subjects with diabetes mellitus.
* Subjects receiving hormone replacement or glucocorticoids.
* Subjects receiving long-term warfarin.
* Subjects suffering from significant systemic diseases, or illnesses that interfere with pituitary-gonadal functions.
* Subjects with a progressive or degenerative neurological disorder.
* Subjects who are unable to take their medication reliably.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2004-11; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Fasting insulin/glucose ratio | 12 months

SECONDARY OUTCOMES:
Number of subjects with above normal upper limit(s) of: insulin level | 12 months
testosterone | 12 months
low-density lipoprotein (LDL) cholesterol | 12 months
luteinizing hormone (LH)/follicle stimulating hormone (FSH) ratio | 12 months
dehydroepiandrosterone (DHEA) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kwan, FHKAM, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - United Christian Hospital, Kowloon
  - Prince of Wales Hospital, Shatin